CLINICAL TRIAL: NCT03719313
Title: A Phase 3, Matrix Design, Partially Double-Blind, Randomized Study of the Efficacy and Safety of 50 mg Lonafarnib/100 mg Ritonavir BID With and Without 180 mcg PEG IFN-alfa-2a for 48 Weeks Compared With PEG IFN-alfa-2a Monotherapy and Placebo Treatment in Patients Chronically Infected With Hepatitis Delta Virus Being Maintained on Anti-HBV Nucleos(t)Ide Therapy (D-LIVR)
Brief Title: Study of the Efficacy and Safety of Lonafarnib / Ritonavir With and Without Pegylated Interferon -Alfa-2a
Acronym: D-LIVR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EIG-LNF-011
Record Dates: First submitted 2018-10-18; First posted 2018-10-25 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis Delta Virus
MeSH Terms: conditions — Hepatitis D | interventions — lonafarnib; Ritonavir; peginterferon alfa-2a

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Lonafarnib 50 mg BID + Ritonavir 100 mg BID
  Interventions: Drug: Lonafarnib; Drug: Ritonavir
- Group 2 (Experimental): Lonafarnib 50 mg BID + Ritonavir 100 mg BID + PEG IFN alfa-2a 180 mcg QW
  Interventions: Drug: Lonafarnib; Drug: Ritonavir; Drug: PEG IFN-alfa-2a
- Group 3 (Active Comparator): placebo Lonafarnib + placebo Ritonavir + PEG IFN-alfa-2a 180 mcg QW
  Interventions: Drug: PEG IFN-alfa-2a; Drug: Placebo Lonafarnib; Drug: Placebo Ritonavir
- Group 4 (Placebo Comparator): placebo Lonafarnib + placebo Ritonavir
  Interventions: Drug: Placebo Lonafarnib; Drug: Placebo Ritonavir

INTERVENTIONS:
Drug: Lonafarnib — Lonafarnib (LNF) 50 mg BID
  Other Names: EBP994; Sarasar; LNF
  Arms: Group 1; Group 2
Drug: Ritonavir — Ritonavir (RTV) 100 mg BID
  Other Names: Norvir; RTV
  Arms: Group 1; Group 2
Drug: PEG IFN-alfa-2a — PEG IFN alfa-2a 180 mcg QW
  Other Names: Pegasys; pegylated interferon-alfa
  Arms: Group 2; Group 3
Drug: Placebo Lonafarnib — Placebo
  Arms: Group 3; Group 4
Drug: Placebo Ritonavir — Placebo
  Arms: Group 3; Group 4

SUMMARY:
Two LNF-containing regimens will be evaluated in the D-LIVR Phase 3 study: (1) LNF/RTV/PEG IFN-alfa-2a and (2) LNF/RTV. Each of these arms will have efficacy endpoints that measure clinical benefit with regard to viral suppression and alanine aminotransferase (ALT) normalization. For each LNF-containing regimen, a composite endpoint of EOT (48 weeks) virologic response and ALT normalization will be used. Virologic response will be defined as a 2 log10 IU/mL reduction from baseline.

DETAILED DESCRIPTION:
This partially double-blind, randomized study will employ a matrix (factorial) design to evaluate the efficacy and safety of LNF 50 mg/RTV 100 mg twice per day (BID) with and without PEG IFN-alfa-2a 180 mcg once-weekly (QW) for 48 weeks compared to no treatment (placebo LNF and placebo RTV) in patients chronically infected with hepatitis delta virus (HDV) and receiving anti-HBV (hepatitis B virus) nucleos(t)ide maintenance therapy.

Approximately 400 patients will be randomized with an allocation ratio of 7:5:2:2 All patients will receive/maintain background anti-HBV nucleos(t)ide therapy with entecavir or tenofovir for at least 12 weeks prior to initiating study therapy.

All patients who complete 48 weeks of treatment will have a liver biopsy for histology assessment at EOT and will be followed for an additional 24 weeks off study treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HDV infection for at least 6 months in duration, documented by a positive HDV antibody test and HDV RNA ≥ 500 IU/mL.

   Note: All genotypes of HDV permitted.
2. Demonstrable suppression of HBV DNA following at least 12 weeks of anti-HBV nucleos(t)ide treatment with entecavir or tenofovir prior to initiating therapy.
3. Serum ALT > 1.3 x upper limit of the normal range (ULN) and < 10 x ULN.
4. Baseline liver biopsy demonstrating evidence of chronic hepatitis.
5. ECGs demonstrating no acute ischemia or clinically significant abnormality.
6. Normal dilated retinal examination.

Exclusion Criteria:

General Exclusions

1. Previous use of LNF within 12 months.
2. Current or previous history of decompensated liver disease.
3. Co-infected with human immunodeficiency virus or hepatitis C virus (HCV) by detectable HIV RNA and HCV RNA, respectively.
4. Evidence of significant portal hypertension.
5. Current evidence or history of ascites requiring diuretics or paracentesis, or hepatic encephalopathy.
6. History of hepatocellular carcinoma.
7. Patients with any of the following:

   * Current eating disorder
   * Evidence of alcohol substance use disorder.
   * Drug abuse within the previous 6 months before screening.
8. Prior history or current evidence of any of the following:

   * Immunologically mediated disease,
   * Retinal disorder or clinically relevant ophthalmic disorder,
   * Any malignancy within 5 years before screening,
   * Cardiomyopathy or significant ischemic cardiac or cerebrovascular disease,
   * Chronic pulmonary disease,
   * Pancreatitis or colitis,
   * Severe or uncontrolled psychiatric disorder.
9. Other significant medical condition that may require intervention during the study.
10. Any condition that may impact proper absorption.
11. Therapy with an immunomodulatory agent, IFN-α (eg, IFN alfa-2a or IFN-alfa-2b, or pegylated IFN-alfa-2a or alfa 2b), cytotoxic agent, or chronic systemic corticosteroids within 12 months of screening.
12. Use of heparin or warfarin.
13. Systemic antibiotics, antifungals, or antivirals for treatment of active infection other than HBV.
14. Receipt of systemic immunosuppressive therapy.
15. History or evidence for any intolerance or hypersensitivity to LNF, RTV, PEG IFN-alfa-2a, tenofovir or entecavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
To compare the composite virologic and biochemical response rate at end-of-treatment (EOT) in patients who receive LNF 50 mg/RTV 100 mg BID vs patients who receive placebo. | 48 weeks
To compare the composite virologic and biochemical response rate at EOT in patients who receive LNF 50 mg/RTV 100 mg BID with PEG IFN-alfa-2a 180 mcg QW vs patients who receive placebo. | 48 weeks

SECONDARY OUTCOMES:
To compare the histologic response rate at EOT in patients who receive LNF 50 mg/RTV 100 mg BID vs patients who receive placebo. | 48 weeks
To compare the histologic response rate at EOT in patients who receive LNF 50 mg/RTV 100 mg BID with PEG IFN-alfa-2a 180 mcg QW vs patients who receive placebo. | 48 weeks
To evaluate the health-related quality of life (HRQL) over a 48-week treatment period in patients who receive LNF 50 mg/RTV 100 mg BID vs placebo. | 48 weeks
To evaluate the HRQL over a 48-week treatment period in patients who receive LNF 50 mg/RTV 100 mg BID/PEG IFN-alfa-2a 180 mcg QW vs placebo. | 48 weeks
To evaluate the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] over a 48-week treatment period in patients who receive LNF 50 mg/RTV 100 mg BID vs placebo. | 48 weeks
To evaluate the Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] over a 48-week treatment period in patients who receive LNF 50 mg/RTV 100 mg BID/PEG IFN-alfa-2a 180 mcg QW vs placebo. | 48 weeks

CONTACTS AND LOCATIONS:
Locations (116):
- United States (18):
  - UCSF Fresno, Fresno, California
  - Ruane Clinical Research Group Inc., Los Angeles, California
  - Asia Pacific Liver Center, Los Angeles, California
  - Stanford University, Palo Alto, California
  - University of California Davis Health System, Sacramento, California
  - Kaiser Permanente Medical Center Sacramento, Sacramento, California
  - Yale University Medical Center, New Haven, Connecticut
  - University of Miami Schiff Center for Liver Disease, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - National Institutes of Health, Bethesda, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mt. Sinai Hospital, New York, New York
  - NYU Langone Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Central Sooner Research, Norman, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
- Belgium (5):
  - ZNA Stuivenberg, Antwerp
  - C.H.U. Brugmann, Brussels
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU Sart Tilman, Liège
- Bulgaria (4):
  - Acibadem City Clinic Tokuda Hospital Ead, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University Health Network, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - McGill University Health Centre/Glen Site / Royal Victoria Hospital, Montreal, Quebec
- France (8):
  - CHU Nice - Hôpital de l'Archet 2, Nice, Alpes Maritimes
  - CHU Strasbourg - Hôpital Hautepierre, Strasbourg, Bas Rhin
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hôpital Beaujon, Clichy, Hauts De Seine
  - CHU de Grenoble - Hôpital Nord, La Tronche, Isere
  - Centre Hospitalier de la Croix Rousse, Lyon, Rhone
  - Hôpital Jean Verdier, Bondy, Seine Saint Denis
  - Hôpital Paul Brousse, Villejuif, Val De Marne
- Germany (8):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Goethe Universität Frankfurt Am Main, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Zentrum für Infektiologie Berlin Prenzlauer Berg GmbH, Berlin
  - Charite - Campus Virchow-Klinikum, Berlin
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
- General Hospital of Athens Laiko, Athens, Greece
- Israel (8):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam Health Care Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
- Italy (13):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Foggia, Foggia
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan
  - Universita di Modena e Reggio Emilia. Nuovo Ospedale civil, Modena
  - Azienda Ospedaliera Universitaria "Federico II", Napoli
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Roma
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Moldova (2):
  - ISMP Spitalul Clinic Republican "Timofei Mosneaga", Chisinau
  - Rtl Sm Srl, Chisinau
- The Liver Center, Ulaanbaatar, Mongolia
- Auckland City Hospital, Grafton, New Zealand
- The Aga Khan University, Karachi, Pakistan
- Romania (6):
  - S.C MedLife S.A, Bucharest
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Bucharest
  - Institutul National de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Fundatia "Dr. Victor Babes", Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
- Russia (11):
  - Clinic of the Ministry of health of the South Ural state medical UNIVERSITY Russia, 2 infectious diseases Department., Chelyabinsk
  - Krasnodar specialized clinical infectious diseases hospital, Krasnodar
  - Modern Medicine Clinic, LLC, Moscow
  - H-Clinic, LLC, Moscow
  - National medical research center Phthisiopulmonology and infectious diseases of the Ministry of health of the Russian Federation, Moscow
  - Healthy Family, LLC, Novosibirsk
  - Clinica UZI 4D, LLC, Pyatigorsk
  - Medical University "Reaviz", Samara
  - Hepatolog, LLC, Samara
  - State Budgetary Educational Institution of Higher Profesional Education "Stavropol State Medical University" of MoH, Stavropol
  - Office for treatment of patients with viral hepatitis GBU Sakha (Yakutia) "Yakut Republican clinical hospital", Yakutsk
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Falu Lasarett, Falun
  - Karolinska Universitetssjukhuset Huddinge, Huddinge
  - Skånes Universitetssjukhus, Malmo
- Inselspital Bern, Hepatologie, Bauchzentrum, INO- A, Ms. Kathrin Husi, Bern, Switzerland
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Chia-Yi Christian Hospital, Chia-Yi City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Linkou, Taoyuan
- Turkey (Türkiye) (3):
  - Dicle University, Medical Faculty, Diyarbakır
  - Koc University Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
- Ukraine (7):
  - Hospital of the state institution "National Institute of Therapy named after L.T. Maloi of the National Academy of Medical Sciences of Ukraine", Kharkiv
  - Medical Center "Harmony of Beauty", LLC, Kyiv
  - Medical Center 'Ok!Clinic+' of International Institute of Clinical Research LLC, Kyiv
  - Medical Center "Preventclinic", LLC, Kyiv
  - Municipal Enterprise "Poltava Regional Clinical Infectious Hospital of Poltava Regional Council", Poltava
  - University Hospital of Sumy State University, Sumy
  - Municipal non-profit enterprise " Vinnytsia city clinical hospital No. 1", Vinnytsia
- United Kingdom (2):
  - Royal London Hospital, London, Greater London
  - Gartnavel General Hospital, Glasgow, Strathclyde

REFERENCES:
- [Derived] Asselah T, Rizzetto M. Hepatitis D Virus Infection. N Engl J Med. 2023 Jul 6;389(1):58-70. doi: 10.1056/NEJMra2212151. No abstract available. PMID 37407002